CLINICAL TRIAL: NCT02342873
Title: A Randomized Comparison of Nerve Stimulator-guided and Ultrasound-guided Interscalene Block for Shoulder Surgery
Brief Title: Nerve Stimulator Versus Ultrasound-guided Interscalene Block for Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cheju Halla General Hospital (Other)
Responsible Party: Principal Investigator, Chunwoo Yang, staff anesthesiologist, Cheju Halla General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: inter2
Record Dates: First submitted 2014-12-11; First posted 2015-01-21 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Pain
Keywords: ultrasound; nerve stimulator
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NS-guided interscalene block (Active Comparator): NS-guided interscalene block is performed using 20 ml of 0.75% ropivacaine.
  Interventions: Procedure: NS-guided interscalene block
- US-guided interscalene block (Experimental): US-guided interscalene block is performed using 20 ml of 0.75% ropivacaine.
  Interventions: Procedure: US-guided interscalene block

INTERVENTIONS:
Procedure: NS-guided interscalene block — Patients received a standard single injection interscalene block using the modified lateral approach of Borgeat. The interscalene brachial plexus was identified using an insulated needle connected to a nerve stimulator. An insulated needle attached to a nerve stimulator was used to identify the brachial plexus. Placement of the needle was considered adequate if the deltoid, triceps, pectoralis, or biceps muscle motor response was still present at 0.2 - 0.5mA. Ropivacine 0.75% 20ml was used.
  Arms: NS-guided interscalene block
Procedure: US-guided interscalene block — Interscalene block is performed under ultrasound guidance. Linear probe is placed on the ipsilateral interscalene groove visualizing the brachial plexus located between anterior and middle scalene muscles. Using in-plane technique, an insulated needle is advanced into the brachial plexus sheath, into which 20 ml of 0.75% ropivacaine is injected
  Arms: US-guided interscalene block

SUMMARY:
The investigators compared the postoperative analgesia of nerve stimulator-guided and ultrasound-guided interscalene block after shoulder surgery.

DETAILED DESCRIPTION:
Ultrasound (US)-guided peripheral nerve block has increased in popularity. It has many advantages such as improved success rate, faster onset time, fewer needle passes, shorter performance time, and reduced procedural pain and vascular puncture. However, there is no information about postoperative analgesia.

Therefore, the investigators tested whether nerve stimulator (NS) - guided interscalene block was inferior to ultrasound-guided block in terms of duration of postoperative analgesia for shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical class I - III patients scheduled to undergo shoulder surgery

Exclusion Criteria:

* coagulopathy, severe pulmonary disease, neuropathy, contralateral diaphragmatic paresis, allergy to study medications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
duration of postoperative analgesia | at 24h after surgery
  time from completion of local anesthetic injection until the first request for an analgesic

SECONDARY OUTCOMES:
onset time (complete block of sensory and motor nerve) | until 30min after completion of local anesthetic
  complete block of sensory and motor nerve
patient discomfort (pain score (0 -10) during the procedure) | at 30 min after block placement
  pain score (0 -10) during the procedure
block performance time (the time between the block needle insertion and needle withdrawal) | at 30 min after block placement
  the time between the block needle insertion and needle withdrawal.
The number of needle redirections | at 30 min after block placement
  either forward or backward movement of needle at least 1 cm or more
paresthesia (presence of paresthesia during the procedure) | at 30 min after block placement
  presence of paresthesia during the procedure
motor block of hand | at 30 min after block placement
  degree of motor block in the operated hand
paresthesia of hand | at 30 min after block placement
  presence of paresthesia in the operated hand
Supplemental analgesia | at 24h after surgery
Pain score | at 24h after surgery
  numerical rating scale (0 - 10)
Patient satisfaction | at 24h after surgery
  Patient satisfaction was evaluated using a two-point score: 1, satisfactory (if necessary, I would have the same anesthetic technique); and 2, unsatisfactory (different anesthetic technique).

CONTACTS AND LOCATIONS:
Overall Officials: Chunwoo Yang, MD, Principal Investigator — Dep. of anesthesia and pain medicine, Cheju Halla General Hospital
Locations (1):
- Cheju Halla General Hopsital, Jeju City, Jeju Special Governing Province, South Korea

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Choi S, McCartney CJ. Evidence Base for the Use of Ultrasound for Upper Extremity Blocks: 2014 Update. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):242-50. doi: 10.1097/AAP.0000000000000155. PMID 25376973
- [Result] Koscielniak-Nielsen ZJ. Ultrasound-guided peripheral nerve blocks: what are the benefits? Acta Anaesthesiol Scand. 2008 Jul;52(6):727-37. doi: 10.1111/j.1399-6576.2008.01666.x. Epub 2008 May 12. PMID 18477070